CLINICAL TRIAL: NCT03974204
Title: Benefit of Analyzing Exosomes in the Cerebrospinal Fluid During the Medical Care of Breast Cancer Patients With Suspicion of Leptomeningeal Metastasis.
Brief Title: Analyses of Exosomes in the Cerebrospinal Fluid for Breast Cancer Patients With Suspicion of Leptomeningeal Metastasis.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Modification of the care habits. We believe today that we are no longer able to carry out this study as initially described.
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Exo-LCR; 2018-A02358-47 (Other: N°ID RCB)
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer; Leptomeningeal Metastasis
Keywords: Cerebrospinal fluid; Proteomic profile
MeSH Terms: conditions — Breast Neoplasms; Meningeal Carcinomatosis | interventions — Probability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cerebrospinal fluid and Blood sample collection (Experimental): Collection of cerebrospinal fluid and blood samples:
  * At initial diagnostic assessment;
  * 1 month and 3 months after initial diagnostic assessment, for patients classified "possible", "probable" or "confirmed" according to EANO-ESMO classification, leading to specific leptomeningeal metastase treatment;
  * In case of symptoms leading to leptomeningeal metastase suspicion and at least 3 months after diagnostic assessment, for patients classified "lack of evidence" according to EANO-ESMO classification.
  Interventions: Procedure: Cerebrospinal fluid and blood sample collection at the initial diagnostic assessment; Procedure: Cerebrospinal fluid and blood sample collection if conclusions of initial diagnostic assessment are "Lack of evidence" according to EANO-ESMO classification; Procedure: Cerebrospinal fluid and blood sample collection if conclusions of initial diagnostic assessment are "confirmed", "probable" or "possible", leading to leptomeningeal metastase specific treatment

INTERVENTIONS:
Procedure: Cerebrospinal fluid and blood sample collection at the initial diagnostic assessment — At the initial diagnostic assessment, 3mL of cerebrospinal fluid and 10 ml of blood sample will be collected in order to determine the proteomic profile. Cerebrospinal fluid will be collected during a lumbar puncture aiming to diagnose leptomeningeal metastases.
Procedure: Cerebrospinal fluid and blood sample collection if conclusions of initial diagnostic assessment are "Lack of evidence" according to EANO-ESMO classification — 3mL of cerebrospinal fluid and 10 ml of blood sample will be collected:
  * When suspected metastatic meningitis symptoms arise and
  * at least 3 months after the initial diagnostic assessment, In order to determine the proteomic profile. Cerebrospinal fluid will be collected during a lumbar puncture aiming to diagnose leptomeningeal metastases.
Procedure: Cerebrospinal fluid and blood sample collection if conclusions of initial diagnostic assessment are "confirmed", "probable" or "possible", leading to leptomeningeal metastase specific treatment — 3mL of cerebrospinal fluid and 10 ml of blood sample will be collected:
  * 1 month after the beginning of the specific treatment,
  * 3 months after the beginning of the specific treatment. Cerebrospinal fluid will be collected during a lumbar puncture aiming to assess treatment response or at intrathecal injection of treatment.

SUMMARY:
This is a multicenter, interventional, prospective study among breast cancer patients with a suspicion of metastatic meningitis. The current study aims to assess the use of proteomic profile issued from cerebrospinal fluid microvesicles for diagnosis of leptomeningeal metastases.

DETAILED DESCRIPTION:
The aim of this study is to describe the association between the initial proteomic profile issued from cerebrospinal fluid microvesicles and the initial cytological analysis of the cerebrospinal fluid in breast cancer patients with a suspicion of metastatic meningitis.

Other objectives of the study include:

* Describing the association between the initial proteomic profile and:

  * the histological types and hormonal receptors status of the breast cancer,
  * the likelihood of leptomeningeal metastasis according to the EANO-ESMO classification (Lack of evidence / possible / probable / confirmed) ,
  * the likelihood of leptomeningeal metastasis according to the EANO-ESMO classification, combined with histological type and hormonal receptors status.
* Evaluate the prognostic value of the proteomic profiling for overall survival, according to the EANO-ESMO classification and other known prognosis factors, in patients classified "possible", "probable" or "confirmed" leading to leptomeningeal metastases specific treatment,
* Evaluate the impact of the evolution of the proteomic profile a month after the start of this treatment on the overall survival, in patients with leptomeningeal metastases specific treatment,
* Evaluate the association between the proteomic profile and the EANO-ESMO classification at least 3 months after the initial EANO-ESMO classification,
* Evaluate the evolution of the proteomic profile 3 months after the initial EANO-ESMO classification, in patients initially classified "lack of evidence", broadly and according to the evolution of cytology, the administered treatments and to the EANO-ESMO response if applicable,
* Compare the proteomic profiles issued from cerebrospinal fluid and blood

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven breast cancer
* Patient with suspected metastatic leptomeningitis
* Age ≥ 18 years
* Patient covered by the French social security regime
* Signed written informed consent

Exclusion Criteria:

* History of cancer other than the one being treated
* Contraindication to carrying out the lumbar puncture or cerebrospinal MRI
* Pregnant or breastfeeding patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Proteomic profiles issued from cerebrospinal fluid at diagnosis | Up to 1 week
  Proteomic profile will be obtained by bioinformatic analysis of cerebrospinal fluid.
Cytology of cerebrospinal fluid at diagnosis | Up to 1 week
  Results of cytological analysis of cerebrospinal fluid will be "Positive", "negative", "equivocal".

SECONDARY OUTCOMES:
Proteomic profiles issued from cerebrospinal fluid | Up to 3 months
  Proteomic profile will be obtained by bioinformatic analysis of cerebrospinal fluid:
  * 1 month and 3 month after the start of a specific treatment of the leptomeningeal metastasis, if applicable,
  * 3 months after the initial diagnosis of leptomeningeal metastasis if the likehood of leptomeningeal metastasis is "lack of evidence".
Histological subtype | Before registration in study
  Histological subtype will be subdivised as invasive ductal breast carcinoma, invasive lobular breast carcinoma, other brest carcinoma.
Hormonal receptors status | Before registration in study
  Hormonal receptors status will be subdivised as:
  * Positive hormonal receptors / Positive HER2
  * Positive hormonal receptors / Negative HER2
  * Negative hormonal receptors / Positive HER2
  * Triple negative
Likehood of leptomeningeal metastasis according to the EANO-ESMO classification. | Up to 3 months after the intial diagnosis
  EANO-ESMO classification is obtained by searching clinical symptoms, cancer cells in the cerebrospinal fluid (obtained by lumbar puncture), signs in RMI. The likehood of leptomeningeal metastasis is:
  * Lack of evidence,
  * Possible,
  * Probable,
  * Confirmed.
Overall survival | Time from date of registration to date of death regardless of the cause, assessed up to 1 year
  Overall survival is defined as time from date of registration to date of death regardless of the cause.
Proteomic profiles issued from blood | Up to 3 months after the intial diagnosis
  Proteomic profile will be obtained by bioinformatic analysis of blood.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie LE RHUN, MD, Principal Investigator — Centre Oscar Lambret
Locations (2):
- France (2):
  - Centre Hospitalier Régional Universitaire de Lille, Lille, Hauts-de-France
  - Centre Oscar Lambret, Lille, Hauts-de-France